CLINICAL TRIAL: NCT01950637
Title: GAPP 2 Survey: Global Attitudes of Patients and Physicians in Insulin Therapy for Type 2 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GAPP2; U1111-1136-2536 (Other: WHO)
Record Dates: First submitted 2013-09-23; First posted 2013-09-25 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with type 2 diabetes mellitus (T2DM)
  Interventions: Behavioral: No treatment given
- Healthcare professionals (HCPs)
  Interventions: Behavioral: survey

INTERVENTIONS:
Behavioral: No treatment given — Completion of 90-item online questionnaire.
  Groups: Patients with type 2 diabetes mellitus (T2DM)
Behavioral: survey — Completion of 58-item online questionnarie.
  Groups: Healthcare professionals (HCPs)

SUMMARY:
This study is conducted Asia, Europe and North America. The aim of this study is to describe insulin therapy adherence and the burden of non-adherence on patient functioning, well-being and diabetes management.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS WITH T2DM:
* Diagnosed with type 2 diabetes by a healthcare professional
* Currently being treated with insulin medication, excluding premix insulin treatment
* Age at least 40 years
* Diagnosed as having type 2 diabetes over the age of 40
* HCPs:
* Primary care physician, diabetes specialist (diabetologist/endocrinologist) or diabetes specialist nurse/diabetes nurse educator
* Have a minimum of 2 years experience within current speciality
* See a minimum of 20 type 2 diabetes patients per month (40 for diabetes specialists), of which at least 10 per month must be on modern (analogue) inulins

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Insulin treated patients with type 2 diabetes, and HCPs involved in the treatment, management of diabetes and care of patients with type 2 diabetes.
Sampling Method: Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Basal insulin dosing irregularities: frequency of missed doses, mistimed doses, or reduced doses (patient questionnaire) | In the past 30 days prior to the day when responding to the online questionnaire
Level of patient dosing irregularity: missed, mistimed and reduced dose (HCP questionnaire) | Day 1 (when responding to the online questionnaire)

SECONDARY OUTCOMES:
Incidence of intentional dosing irregularities and reasons for this behaviour | Day 1 (when responding to the online questionnaire)
Impact of dosing irregularity on functional well-being | Day 1 (when responding to the online questionnaire)
Frequency of self-treated hypoglycaemia | In the past 30 days prior to the day when responding to the online questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (6):
- Novo Nordisk Investigational Site, Princeton, New Jersey, United States
- Novo Nordisk Investigational Site, Mississauga, Canada
- Novo Nordisk Investigational Site, Copenhagen S, Denmark
- Novo Nordisk Investigational Site, Mainz, Germany
- Novo Nordisk Investigational Site, Tokyo, Japan
- Novo Nordisk Investigational Site, Crawley, United Kingdom

REFERENCES:
- [Result] Brod M, Rana A, Barnett AH. Impact of self-treated hypoglycaemia in type 2 diabetes: a multinational survey in patients and physicians. Curr Med Res Opin. 2012 Dec;28(12):1947-58. doi: 10.1185/03007995.2012.743457. Epub 2012 Nov 14. PMID 23150950
- [Result] Brod M, Rana A, Barnett AH. Adherence patterns in patients with type 2 diabetes on basal insulin analogues: missed, mistimed and reduced doses. Curr Med Res Opin. 2012 Dec;28(12):1933-46. doi: 10.1185/03007995.2012.743458. Epub 2012 Nov 14. PMID 23150949
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com